CLINICAL TRIAL: NCT06725563
Title: Endoscopically Placed Lumen-Apposing Metal Stents as a Safe Alternative to Surgery for the Treatment of Symptomatic Intestinal Strictures in Individuals With Inflammatory Bowel Disease
Brief Title: Endoscopically Placed Lumen-Apposing Metal Stents for the Treatment of Symptomatic Intestinal Strictures in Individuals With Inflammatory Bowel Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRRF ID: 5849
Record Dates: First submitted 2024-05-28; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Inflammatory Bowel Diseases; Stricture; Bowel
MeSH Terms: conditions — Inflammatory Bowel Diseases; Constriction, Pathologic

STUDY DESIGN:
Intervention Model Description: Participants will receive lumen-apposing metal stents (LAMS) as a treatment for IBD-related strictures. The size of the stent used will depend on the length of the stricture. All LAMS placements are part of a single arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endoscopically placed lumen-apposing metal stents for the treatment of IBD-strictures (Experimental): Individuals will receive endoscopic lumen-apposing metal stents. The specific size of the stent used will depend on the length of the stricture. All LAMS placements are part of one arm.
  Interventions: Procedure: Endoscopically placed lumen-apposing metal stents for the treatment of IBD-strictures

INTERVENTIONS:
Procedure: Endoscopically placed lumen-apposing metal stents for the treatment of IBD-strictures — We will apply standard procedures for endoluminal stenting. A therapeutic colonoscope will be advanced through the bowel up until the stricture. A guidewire will be passed through the lumen at the stricture site. LAMS will be used for strictures <6cm, with stents ranging in size from 10-16mm in diameter and up to 60mm in length. The stent will be deployed across the stricture with the assistance of endoscopic and fluoroscopic imaging. Individuals will undergo a repeat colonoscopy in 1-3 months to remove the stent.

SUMMARY:
This is a single-center prospective pilot study in patients with symptomatic partially obstructing intestinal strictures without severe active inflammation or penetrating complications, evaluating the use of LAMS with respect to symptom and quality of life improvement and the development of stent-related complications.

DETAILED DESCRIPTION:
This will be a prospective case series study in ~20 IBD patients with symptomatic partially-obstructing intestinal strictures < 6 cm in length without severe active inflammation (large or deep ulcers at distal entrance or moderate-severe friability or severe inflammatory changes in the stricture on radiographic imaging, at the discretion of the referring IBD physician or treating therapeutic endoscopist) or penetrating complications (pre-stenotic fistula or intra-abdominal phlegmon or abscess), evaluating the use of LAMS with respect to symptom and quality of life improvement and the development of stent-related complications.

The objective of this project is to evaluate the safety and efficacy of LAMS for the treatment of short segment, symptomatic, IBD-related strictures.

The hope is that positive results from this pilot study will provide sufficient rationale to trigger a larger scale multicenter study to fully assess the efficacy of endoscopic stenting for IBD-related strictures.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Established Diagnosis of inflammatory bowel disease
* Symptomatic, single, fibrostenotic or anastomotic stricture <6 cm in length without severe active inflammation, pre-stenotic intestinal fistula or penetrating complication, and within reach of the adult colonoscope (colon or terminal ileum)
* Ability to accurately gauge stricture length with imaging and safely deploy the stent using conventional fluoroscopic techniques
* Able to provide informed consent

Exclusion Criteria:

* More than one intestinal stricture
* Stricture out of reach of standard adult colonoscope
* High-grade stricture (complete or near complete bowel obstruction
* Severe active inflammation in the stricture or associated penetrating complication, including fistula, inflammatory phlegmon or abscess
* Contraindications for endoscopic therapy, including:
* Complete Bowel obstruction
* Severe cardiorespiratory comorbidity
* Unable to tolerate sedation or anesthesia
* Non-reversible coagulopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical success | 12-months following stent removal
  defined as persistent improvement of obstructive symptoms and establishment of adequate oral caloric intake at 12 months following stent removal, measured using quality of life pre- and post-endoscopic stenting measured using short inflammatory bowel disease questionnaire (SIBDQ), pre- and post-stenting nutritional/health outcomes measured using Saskatchewan IBD-Nutrition Risk (SaskIBD-NR Tool)

SECONDARY OUTCOMES:
Technical success | 1-3 months
  defined as successful deployment of the stent without stent-related complications, including stent migration or perforation by the time of stent removal
Patient satisfaction | 12 months
  Endoscopic stenting patient satisfaction measured using a decision regret form
Incidence of adverse events | 12 months
  Incidence of post procedure adverse events (stent migration, abdominal pain, perforation, infection, bleeding)

CONTACTS AND LOCATIONS:
Overall Officials: Avijit Chatterjee, MD, MSc., Principal Investigator — Ottawa Hospital Research Institute

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared.

REFERENCES:
- [Background] Coward S, Benchimol EI, Kuenzig ME, Windsor JW, Bernstein CN, Bitton A, Jones JL, Lee K, Murthy SK, Targownik LE, Pena-Sanchez JN, Rohatinsky N, Ghandeharian S, Im JHB, Davis T, Weinstein J, Goddard Q, Bennett J, Caplan L, Bergevin M, Yang XY, Mason K, Sanderson R, Brass C, Kaplan GG. The 2023 Impact of Inflammatory Bowel Disease in Canada: Epidemiology of IBD. J Can Assoc Gastroenterol. 2023 Sep 5;6(Suppl 2):S9-S15. doi: 10.1093/jcag/gwad004. eCollection 2023 Sep. PMID 37674492
- [Background] Mitropoulou MA, Fradelos EC, Lee KY, Malli F, Tsaras K, Christodoulou NG, Papathanasiou IV. Quality of Life in Patients With Inflammatory Bowel Disease: Importance of Psychological Symptoms. Cureus. 2022 Aug 28;14(8):e28502. doi: 10.7759/cureus.28502. eCollection 2022 Aug. PMID 36185946
- [Background] Nasr S, Dahmani W, Jaziri H, Hammami A, Slama AB, Ameur WB, Elleuch N, Ksiaa M, Jmaa A. Exploring work productivity loss in patients with inflammatory bowel disease. Future Sci OA. 2023 Jun 7;9(8):FSO872. doi: 10.2144/fsoa-2022-0034. eCollection 2023 Sep. PMID 37621842
- [Background] Shen B. Principles, Preparation, Indications, Precaution, and Damage Control of Endoscopic Therapy in Inflammatory Bowel Disease. Gastrointest Endosc Clin N Am. 2022 Oct;32(4):597-614. doi: 10.1016/j.giec.2022.05.005. Epub 2022 Sep 7. PMID 36202505
- [Background] Kuenzig ME, Benchimol EI, Lee L, Targownik LE, Singh H, Kaplan GG, Bernstein CN, Bitton A, Nguyen GC, Lee K, Cooke-Lauder J, Murthy SK. The Impact of Inflammatory Bowel Disease in Canada 2018: Direct Costs and Health Services Utilization. J Can Assoc Gastroenterol. 2019 Feb;2(Suppl 1):S17-S33. doi: 10.1093/jcag/gwy055. Epub 2018 Nov 2. PMID 31294382
- [Background] Lin V, Gogenur S, Pachler F, Fransgaard T, Gogenur I. Risk Prediction for Complications in Inflammatory Bowel Disease Surgery: External Validation of the American College of Surgeons' National Surgical Quality Improvement Program Surgical Risk Calculator. J Crohns Colitis. 2023 Jan 27;17(1):73-82. doi: 10.1093/ecco-jcc/jjac114. PMID 35973971
- [Background] Wiebe K, Kelley S, Kirsch RE. Revisiting the concept of urgency in surgical prioritization and addressing backlogs in elective surgery provision. CMAJ. 2022 Aug 2;194(29):E1037-E1039. doi: 10.1503/cmaj.220420. No abstract available. PMID 35918085
- [Background] Springer JE, Doumouras AG, Saleh F, Lee J, Amin N, Cadeddu M, Eskicioglu C, Hong D. Drivers of Inpatient Costs After Colorectal Surgery Within a Publicly Funded Healthcare System. Dis Colon Rectum. 2019 Jun;62(6):747-754. doi: 10.1097/DCR.0000000000001309. PMID 31094961
- [Background] Jeong SJ, Park J. Endoscopic Management of Benign Colonic Obstruction and Pseudo-Obstruction. Clin Endosc. 2020 Jan;53(1):18-28. doi: 10.5946/ce.2019.058. Epub 2019 Oct 24. PMID 31645090
- [Background] Jena A, Chandnani S, Jain S, Sharma V, Rathi P. Efficacy of endoscopic over-the-scope clip fixation for preventing migration of self-expandable metal stents: a systematic review and meta-analysis. Surg Endosc. 2023 May;37(5):3410-3418. doi: 10.1007/s00464-023-09893-z. Epub 2023 Jan 30. PMID 36717426
- [Background] Sharma P, McCarty TR, Chhoda A, Costantino A, Loeser C, Muniraj T, Ryou M, Thompson CC. Alternative uses of lumen apposing metal stents. World J Gastroenterol. 2020 Jun 7;26(21):2715-2728. doi: 10.3748/wjg.v26.i21.2715. PMID 32550749
- [Background] Nunez F P, Krugliak Cleveland N, Quera R, Rubin DT. Evolving role of endoscopy in inflammatory bowel disease: Going beyond diagnosis. World J Gastroenterol. 2021 May 28;27(20):2521-2530. doi: 10.3748/wjg.v27.i20.2521. PMID 34092973
- [Background] Chandan S, Dhindsa BS, Khan SR, Deliwala S, Kassab LL, Mohan BP, Chandan OC, Loras C, Shen B, Kochhar GS. Endoscopic Stenting in Crohn's Disease-related Strictures: A Systematic Review and Meta-analysis of Outcomes. Inflamm Bowel Dis. 2023 Jul 5;29(7):1145-1152. doi: 10.1093/ibd/izac153. PMID 35880681
- [Background] Medas R, Ferreira-Silva J, Girotra M, Barakat M, Tabibian JH, Rodrigues-Pinto E. Best Practices in Esophageal, Gastroduodenal, and Colonic Stenting. GE Port J Gastroenterol. 2022 Nov 7;30(Suppl 1):19-34. doi: 10.1159/000527202. eCollection 2023 Sep. PMID 37818397
- [Background] Das R, Singh R, Din S, Lund J, Krishnamoorthy R, Hearing S, Norton B, Williams J, Fraser C, Goddard A, Cole A. Therapeutic resolution of focal, predominantly anastomotic Crohn's disease strictures using removable stents: outcomes from a single-center case series in the United Kingdom. Gastrointest Endosc. 2020 Aug;92(2):344-352. doi: 10.1016/j.gie.2020.01.053. Epub 2020 Feb 18. PMID 32081614
- [Background] Hedenstrom P, Stotzer PO. Endoscopic treatment of Crohn-related strictures with a self-expandable stent compared with balloon dilation: a prospective, randomised, controlled study. BMJ Open Gastroenterol. 2021 Mar;8(1):e000612. doi: 10.1136/bmjgast-2021-000612. PMID 33722805